CLINICAL TRIAL: NCT06534372
Title: Affecting Factors the Incidince of Chronic Pain After Sternotomy
Brief Title: Affecting Factors for Chronic Pain After Sternotomy
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Umut Can Özağar, Principal İnvestigator, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK1-2024-0068
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Surgery; Sternotomy; Pain, Acute; Pain, Chronic
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Sternotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Open cardiac surgery with sternotomy — Factors affecting the occurrence of chronic pain in patients undergoing open cardiac surgery with sternotomy will be investigated.

SUMMARY:
Chronic pain is common complication of surgery procedures. Rates of mortalits is getting lower in cardiac surgery. This situation has brought us to focus morbidity and long term life quality. Previous study show that chronic pain after cardiac surgery is experienced 11-40% patient. Multifactorial causes play a role in chronic pain etiology. The aim of our study is to determine the causes of chronic pain in patients who underwent sternotomy.

DETAILED DESCRIPTION:
Pain can be classified as anatomical, etiological, duration, intensity, and pathophysiological.

Classification according to duration is made according to the duration that the person feels the pain. Here, the classification is basically divided into acute and chronic. Acute pain is usually associated with acute injury or trauma. Chronic pain is defined as pain that continues after the expected period for the tissues to heal. Chronic pain is pain that lasts for 3 months or longer. Various conditions, usually including psychological and ethnic conditions, can affect the type of pain.

More than 2 million people worldwide undergo open heart surgery. Although mortality rates have decreased significantly thanks to advances in anesthesia and surgery, chronic pain after open heart surgery is still a serious problem. The rate of chronic pain varies between 11-40% within 1 year after cardiac surgery. Since open heart surgery is a very common procedure, it affects many people. Therefore; It is important to understand the factors related to the development of chronic pain.

Many risk factors have been identified for chronic pain after coronary artery bypass surgery. These are; female gender, young age, preoperative anxiety, intraoperative opioid use, and intense pain in the first days of the postoperative period. Although there are various retrospective and prospective studies on this subject, these studies are still insufficient and need support in the literature.

In this study, investigators aim to reveal the factors that increase chronic pain after sternotomy, take precautions against these factors and reduce the development of chronic pain.

Chronic pain is a problem that has been increasing in our country as well as all over the world in recent years. Therefore, defining the factors related to pain is very important. In our study, investigators aim to reveal the factors that increase chronic pain after sternotomy. By determining these factors, it will be possible to prevent the development of chronic pain in patients, reduce costs and increase the quality of life of patients. This study does not pose any risk for the patients to be included.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-80
* BMI 18-35 kg/m2
* ASA (American Society of Anesthesiologists) Scoring I-II-III
* Elective open coronary artery bypass graft surgery
* Elective open heart valve surgery
* Patients who will undergo general anesthesia
* Patients who agree to participate in the study and sign a form

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* Patients who do not want to participate in the study
* Patients with advanced organ failure (liver failure, renal failure)
* Patients with chronic pain or chronic opioid use
* Patients with alcohol, substance or drug addiction
* Patients planned for surgery with thoracotomy
* Patients with a history of previous sternotomy (redo)
* Patients with limited cooperation such as dementia, psychiatric disorders
* Pregnant and breastfeeding patients will be excluded from the study.
* Patients who cannot communicate in their native language will be excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the ASA I-II-III risk group, between the ages of 18-80 years, with a BMI between 18-35 kg/m2, who will undergo elective open coronary artery bypass graft surgery, who will undergo elective open heart valve surgery, who will undergo general anesthesia, and who will undergo sternotomy will be included in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Self-leeds assessment of neuropathic symptoms and sign findings in 3rd months. | 3rd postoperative month
  Patients' self-Leeds assessment of neuropathic symptoms and sign (S-LANSS) findings will be evaluated in the 3rd postoperative month. Patients with an S-LANSS score of 12 and above will be diagnosed with chronic neuropathic pain.

SECONDARY OUTCOMES:
Self-leeds assessment of neuropathic symptoms and sign findings at 6th months | 6th postoperative month
  Patients' self-Leeds assessment of neuropathic symptoms and sign (S-LANSS) findings will be evaluated in the 3rd postoperative month. Patients with an S-LANSS score of 12 and above will be diagnosed with chronic neuropathic pain.
Short Form 12 scores in the 3rd month. | 3rd postoperative month
  Short Form 12 scores will be evaluated in the 3rd month to evaluate the quality of life of the patients.
Short Form 12 scores in the 6th month. | 6th postoperative month
  Short Form 12 scores will be evaluated in the 6th month to evaluate the quality of life of the patients.
Acute pain score | Up to postoperative 24 hour
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be made in 1, 2, 12, 24 hour after extubation in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Jülide Ergil, Professor, Study Director — WHO, Turkish Society of Anesthesiology and Reanimation
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Etlik City Hospital, Ankara, Ankara
  - Ankara Etlik City Hospital, Ankara, Yenimahalle

IPD SHARING:
Plan to Share IPD: No